CLINICAL TRIAL: NCT03654248
Title: Randomized Controlled Trial of "Let's Get Organized"; an Intervention Program for Improving Time Management Skills in Adults with Cognitive Limitations
Brief Title: "Let's Get Organized" in Adult Psychiatric/habilitation Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Örebro University, Sweden (Other)
Collaborators: Region Örebro County (Other); Dalarna County Council, Sweden (Other); Uppsala University (Other); Region Gävleborg (Other); State University of New York - Downstate Medical Center (Other); Uppsala County Council, Sweden (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORU 2018/191
Record Dates: First submitted 2018-08-20; First posted 2018-08-31 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2023-03

CONDITIONS: Neurodevelopmental Disorders; Mental Disorder
Keywords: Time management; Group intervention; Executive function
MeSH Terms: conditions — Neurodevelopmental Disorders; Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Let's Get Organized group intervention (Experimental): Group intervention with 10 weekly sessions, each lasting 1,5 hours
  Interventions: Behavioral: Let's Get Organized group intervention
- Individual Occupational Therapy (Active Comparator): Individual intervention lasting 10 weeks
  Interventions: Device: Individual Occupational Therapy

INTERVENTIONS:
Behavioral: Let's Get Organized group intervention — Group intervention aiming to enhance time management, targeted to persons with mental or neurodevelopment disorders. Each group has 6-8 participants and is lead by two trained group leaders. Goal-directed and other learning strategies are used to train effective time management habits such as maintaining a calendar and wearing a watch. Group sessions are structured with PowerPoint presentation and a course manual, an information from the group leaders is intermixed with discussion among the participants and tasks to complete.
  Other Names: LGO
  Arms: Let's Get Organized group intervention
Device: Individual Occupational Therapy — Individual meetings with Occupational Therapist (standard therapy) during a 10-week period. Number of meetings and exact nature of intervention depends on the client's needs and is decided by the treating occupational therapist. Interventions will include prescription or instruction regarding time assistive devices and instructions regarding structure and planning of everyday life.
  Arms: Individual Occupational Therapy

SUMMARY:
This project aims to evaluate and establish evidence for a novel, group-based intervention that can help people with cognitive limitations due to mental or neurodevelopmental disorders to improve their ability to manage time and organize activities. This might provide an important step towards establishing healthy life habits, getting or maintaining employment, and managing family life. Time management is a necessary skill for maintaining healthy life habits and daily occupations in modern society. People with limited cognitive function due to, for example, mental or neurodevelopmental disorders, have documented difficulties in time management, which is also related to issues with self-efficacy. Common interventions for persons with poor time management are time-assistive devices and products, but studies show that these devices alone are not enough to cover these people's needs. Structured training is needed, but there is a lack of structured interventions to enhance time management skills. The intervention program "Let's get organized" (LGO) is a manual-based group intervention aiming to enhance time management, targeted to persons with mental or neurodevelopmental disorders. In a recent feasibility study the LGO showed promising results.

This project aims to evaluate to what extent the LGO intervention is effective in improving time management, and satisfaction with daily occupations. The proposed project is a randomized-controlled trial carried out in ten psychiatric units in Sweden. Participants (n=104) will be randomly assigned to either LGO group intervention or individual Occupational Therapy intervention for ten weeks .The primary outcome of the study is self-reported time management measured by the Assessment of Time Management Skills. Secondary outcomes are occupational balance, self-efficacy, parental competence and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* confirmed or suspected diagnosis of a mental disorder, such as affective disorder or schizophrenia, or neurodevelopment disorder, such as autism spectrum disorder or attention deficit hyperactivity disorder/attention deficit disorder
* self-reported difficulties in time management in daily life to an extent that affects functioning in daily life negatively

Exclusion Criteria:

* intellectual disability

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Assessment of Time Management Skills-Swedish, Time management sub scale at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  11 items, reported as 0-100 ATMS units

SECONDARY OUTCOMES:
Change in Weekly Calendar Planning Activity-Swedish version No of correct appointments at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Performance test of executive functioning. No of correctly entered appointments (range 0-17)
Change in Weekly Calendar Planning Activity Swedish version total time at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Performance test of executive functioning. Total time
Change in Weekly Calendar Planning Activity Swedish version no of strategies at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Performance test of executive functioning. No of strategies used more strategies are better
Change in Weekly Calendar Planning Activity Swedish version rules followed at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Performance test of executive functioning. No of rules followed (range 0-5) More rules followed are better
Change in Weekly Calendar Planning Activity Swedish version efficacy score at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Performance test of executive functioning. Efficacy score (high score is better)
Change in Satisfaction with daily occupations and occupational balance (SDO-OB) activity score at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  No of activities (range 0-17, higher scores are better)
Change in Satisfaction with daily occupations and occupational balance (SDO-OB) satisfaction score at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Satisfaction score (range 13-91, higher scores are better)
Change in Global satisfaction score at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Global satisfaction score (range 1-5, lower scores are better)
Change in Satisfaction with daily occupations and occupational balance (SDO-OB) occupational balance at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Occupational balance (nominal data)
Change in General Self-Efficacy Scale at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Self-efficacy (range 0-40, higher score is better)
Change in Parental Sense of Competence at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Sense of competence (range 15-90, higher score is better)
Change in EuroQuality of Life - 5 dimensions - 5 levels (EQ-5D-5L) item scores at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  Individual item scores on 5 items scored 1-5
Change in EuroQuality of Life - 5 dimensions - 5 levels (EQ-5D-5L) global score at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  One visual-analogue-scale answer (range 0-100)
Change in Assessment of Time Management Skills-Swedish (ATMS-S), Organization and planning sub scale at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  11 items, reported as 0-100 ATMS units
Change in Assessment of Time Management Skills-Swedish (ATMS-S), Regulation of emotions sub scale at 10 weeks after intervention start and at 24 weeks after intervention start | baseline (pre-intervention), 10 weeks, 24 weeks
  5 items, reported as 0-100 ATMS units
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: depression domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: anger domain | baseline (pre-intervention), 10 weeks, 24 weeks
  1 item, reported as 0-4 points
Change in DSM-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: mania domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: anxiety domain | baseline (pre-intervention), 10 weeks, 24 weeks
  3 items, reported as 0-12 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: somatic symptoms domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in DSM-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: suicidal ideation domain | baseline (pre-intervention), 10 weeks, 24 weeks
  1 items, reported as 0-4 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: psychosis domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: sleep problems domain | baseline (pre-intervention), 10 weeks, 24 weeks
  1 items, reported as 0-4 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: memory domain | baseline (pre-intervention), 10 weeks, 24 weeks
  1 items, reported as 0-4 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: repetitive thoughts and behaviors domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: dissociation domain | baseline (pre-intervention), 10 weeks, 24 weeks
  1 items, reported as 0-4 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: personality functioning domain | baseline (pre-intervention), 10 weeks, 24 weeks
  2 items, reported as 0-8 points
Change in Diagnostic and Statistical Manual of Mental Disorders Manual-5 Self-rated level 1 Cross-Cutting Symptom Measure Adult: substance use domain | baseline (pre-intervention), 10 weeks, 24 weeks
  3 items, reported as 0-12 points
Autism Quotient Short | baseline (pre-intervention), 10 weeks, 24 weeks
  28 items, 28-112 points
Adult Attention Deficit Hyperactivity disorder Self-report Scale | baseline (pre-intervention), 10 weeks, 24 weeks
  18 items, score 1-90

CONTACTS AND LOCATIONS:
Overall Officials: Marie Holmefur, PhD, Principal Investigator — Örebro University, Sweden
Locations (8):
- Sweden (8):
  - Öppenvårdspsykiatrisk mottagning, Falun, Dalarna County
  - Habiliteringscenter Brommaplan vuxna, Habilitering och Hälsa, Region Stockholm, Stockholm
  - Neuropsykiatriska mottagningen, Akademiska sjukhuset, Uppsala
  - Hallsberg psykiatrisk öppenvård, Hallsberg, Örebro County
  - Karlskoga psykiatrisk öppenvård, Karlskoga, Örebro County
  - Lindesberg psykiatrisk öppenvård, Lindesberg, Örebro County
  - USÖ psykiatrisk öppenvård och affektiva enhet, Örebro, Örebro County
  - Vuxenhabiliteringen - Autismteamet, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holmefur M, Roshanay A, White S, Janeslatt G, Vimefall E, Lidstrom-Holmqvist K. Evaluation of the "Let's Get Organized" group intervention to improve time management: protocol for a multi-centre randomised controlled trial. Trials. 2021 Sep 19;22(1):640. doi: 10.1186/s13063-021-05578-x. PMID 34538253